CLINICAL TRIAL: NCT02743806
Title: Entyvio (Vedolizumab IV) Extended Access Program in Ulcerative Colitis and Crohn's Disease
Brief Title: Extended Access Program of Vedolizumab IV in Ulcerative Colitis and Crohn's Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Early Completed - Alternative Source of Drug Available
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vedolizumab-4013; 2016-000678-40 (EudraCT Number); U1111-1180-9339 (Registry Identifier: WHO)
Record Dates: First submitted 2016-04-15; First posted 2016-04-19 (Estimated); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Colitis, Ulcerative; Crohn Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg, IV infusion, once every 8 weeks (Q8W) that maybe reduced to once every 4 weeks (Q4W) based on the investigator's judgment of participant's clinical status and acknowledged by the medical monitor for up to 6 years.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab IV infusion
  Other Names: MLN0002; Entyvio; Kynteles

SUMMARY:
The purpose of this study is to monitor ongoing safety in participants with ulcerative colitis (UC) and Crohn's disease (CD) and to provide access to vedolizumab for qualifying participants who, in the opinion of the investigator, continue to derive benefit from vedolizumab and for whom continued treatment with vedolizumab is desired because there is no other comparable product available or the participant may be expected to develop worsening of disease if they were to modify treatment.

DETAILED DESCRIPTION:
The drug being used in this study is called vedolizumab, which is being used to treat people who have ulcerative colitis or Crohn's disease. This study will monitor ongoing safety in the people who take vedolizumab.

Participants who have successfully completed the participation in qualifying vedolizumab clinical studies will be enrolled and assigned to receive:

• Vedolizumab 300 mg

All participants will receive an intravenous (IV) infusion once every 8 weeks until vedolizumab is available through commercial channels, including reimbursement, for the participant's clinical scenario, or until participant withdrawal, whichever comes first. (Per MM approval, dosing regimen may be modified) This multicenter trial will be conducted worldwide. Participants will make multiple visits to the clinic and a final visit at 18 weeks after receiving the last dose of study infusion of vedolizumab for a safety follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Received vedolizumab (excluding comparator or placebo participants) during participation in a qualifying vedolizumab study.
2. In the opinion of the investigator, the participant is continuing to derive benefit from vedolizumab and continued treatment with vedolizumab is desired because there is no other comparable product available or the participant may be expected to develop worsening of disease if they were to modify treatment.
3. A male participant who is non-sterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 18 weeks after last dose.
4. A female participant of childbearing potential who is sexually active with a non-sterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 18 weeks after last dose.

Exclusion Criteria:

1. For the participant's particular clinical scenario, vedolizumab is currently available to the participant through commercial channels, including reimbursement.
2. Has any clinical condition or prior therapy that, in the opinion of the investigator, would make the participant unsuitable for the study or unable to comply with the dosing requirements or poses a risk to the participant being in the study.
3. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 18 weeks after participating in this study; or intending to donate ova during such time period.
4. If male, the participant intends to donate sperm during the course of this study or for 18 weeks thereafter.
5. Has received a live vaccine in the last 18 weeks or is in need of a live vaccine during the study or up to 18 weeks after the last study dose.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (78):
- Australia (6):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Western Hospital, Footscray, Victoria
  - Cabrini Medical Centre, Malvern, Victoria
  - Box Hill Hospital, Box Hill
  - Royal Brisbane & Women's Hospital, Herston
  - Fiona Stanley Hospital, Murdoch
- Bulgaria (2):
  - Multiprofile Hospital For Active Treatment Ruse, Rousse
  - City Clinic University Multiprofile Hospital for Active Treatment EOOD, Sofia
- Czechia (10):
  - Karlovarska krajska nemocnice a.s., Karlovy Vary, Karlovarsk Kraj
  - Hepato-Gastroenterologie HK, s. r. o., Hradec Králové
  - Oblastni nemocnice Kladno, a.s., Kladno
  - Nemocnice Pardubickeho kraje, a.s. Pardubicka nemocnice, Pardubice
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Institut klinicke a experimentalni mediciny, Prague
  - ISCARE I.V.F. a.s., Prague
  - Nemocnice Strakonice, a.s., Strakonice
  - Nemocnice Tabor, a.s., Tábor
  - Krajska zdravotni, a.s. Masarykova nemocnice v Usti nad Labem, o.z., Ústí nad Labem
- Estonia (2):
  - West Tallinn Central Hospital, Tallinn
  - East Tallinn Central Hospital, Tallinn
- Hungary (14):
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged, Csongrád megye
  - Bekes Megyei Kozponti Korhaz, Békéscsaba
  - Peterfy Sandor utcai Korhaz-Rendelintezet es Baleseti Kozpont, Budapest
  - Semmelweis Egyetem, Budapest
  - Szent Janos Korhaz es Eszak-Budai Egyesitett Korhazak, Budapest
  - Szent Pantaleon Korhaz-Rendelointezet, Dunaújváros
  - Bugat Pal Korhaz, Gyöngyös
  - Bekes Megyei Kozponti Korhaz, Gyula
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Karolina Korhaz Rendelointezet, Mosonmagyaróvár
  - Kanizsai Dorottya Korhaz, Nagykanizsa
  - Pecsi Tudomanyegyetem, Pécs
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- India (5):
  - Owaisi Hospital and Research Centre, Hyderabad, Andhra Pradesh
  - Lakeshore Hospital, Kochi, Kerala
  - KEM Hospital Research Centre, Pune, Maharashtra
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - VGM Hospital Institute of Gastroenterology, Coimbatore, Tamil Nadu
- Italy (2):
  - Policlinico San Donato, San Donato Milanese, Milano
  - Istituto Clinico Humanitas, Rozzano
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- New Zealand (3):
  - Christchurch Hospital, Christchurch, Canterbury
  - Waikato Hospital, Hamilton, Waikato Region
  - Shakespeare Specialist Group, Auckland
- Poland (10):
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - Wojewodzki Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie, Krakow, Lesser Poland Voivodeship
  - Ars Medica, Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne sw. Lukasza, Częstochowa, Silesian Voivodeship
  - SPZOZ Wojewodzki Szpital Zespolony im J Sniadeckiego, Bialystok
  - 10 Wojskowy Szpital Kliniczny z Poliklinika, Bydgoszcz
  - Corpora-Med, Gliwice
  - Centrum Zdrowia Matki, Dziecka i Mlodziezy, Warsaw
  - Centralny Szpital Kliniczny MSW, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Romania (2):
  - Colentina Clinical Hospital, Bucharest
  - Fundeni Clinical Institute, Bucharest
- Russia (6):
  - City Clinical Hospital #24, Moscow
  - Nizhegorodskaya Regional Clinical Hospital n.a. Semashko, Nizhny Novgorod
  - Russian Medical Military Academy n.a. S.M. Kirov, Saint Petersburg
  - Union Clinic, LLC, Saint Petersburg
  - St.Petersburg Multi Field City Hospital #2, Saint Petersburg
  - Medical Company Hepatolog, LLC, Samara
- Military Medical Academy, Belgrade, Serbia
- South Africa (4):
  - CLINRESCO, ARWYP Medical Suites, Johannesburg, Gauteng
  - St Augustines Medical Centre, Durban, KwaZulu-Natal
  - Kingsbury Hospital, Claremont, Western Cape
  - Universitas Hospital, Bloemfontein
- South Korea (6):
  - Yeungnam University Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
  - Kyung Hee University Hospital, Seoul
  - Samsung Medical Center - PPDS, Seoul
  - Asan Medical Center - PPDS, Seoul
- Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi, Istanbul, Turkey (Türkiye)
- Ukraine (2):
  - Medical Clinical Research Center of Medical Center LLC Health Clinic, Vinnytsia, Vinnytsia Oblast
  - Poltava Regional Clinical Hospital n.a. M.V. Skliphosovskyi, Poltava

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Danese S, Subramaniam K, Van Zyl J, Adsul S, Lindner D, Roth J, Vermeire S. Vedolizumab treatment persistence and safety in a 2-year data analysis of an extended access programme. Aliment Pharmacol Ther. 2021 Jan;53(2):265-272. doi: 10.1111/apt.16160. Epub 2020 Nov 18. PMID 33210333
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b60394db2bf003ab4a23d?idFilter=%5B%22Vedolizumab-4013%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 78 investigative sites in Australia, Bulgaria, the Czech Republic, Estonia, Hungary, India, Italy, Republic of Korea, Latvia, Malaysia, New Zealand, Poland, Romania, Russian Federation, Serbia, South Africa, Turkey, and Ukraine from 01 August 2016 to 03 January 2023.
Pre-assignment Details: A total of 331 participants with a diagnosis of ulcerative colitis (UC) or Crohn's disease (CD) who have successfully completed the participation in qualifying vedolizumab clinical studies (C13008 [NCT00790933] and MLN0002-3028 [NCT02425111]) were enrolled in this extended access program (XAP) study to receive vedolizumab 300 mg.
Groups:
- Vedolizumab 300 mg: Vedolizumab 300 mg, intravenous (IV) infusion, once every 8 weeks (Q8W) that maybe reduced to once every 4 weeks (Q4W) based on the investigator's judgment of participant's clinical status and acknowledged by the medical monitor for up to 6 years.
Period: Overall Study
Arm/Group | Vedolizumab 300 mg
Started | 331
Completed | 150
Not Completed | 181
Not completed — Adverse Event | 9
Not completed — Lost to Follow-up | 8
Not completed — Voluntary Withdrawal | 54
Not completed — Study Termination | 65
Not completed — Pregnancy | 6
Not completed — No Longer Clinically Benefiting | 27
Not completed — Reason Not Specified | 12

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) consisted of all participants enrolled in the XAP study, who received at least 1 dose of study drug (i.e., vedolizumab IV treatment), including the dose given at T0 (last vedolizumab dose in the qualifying study).
Groups:
- Vedolizumab 300 mg: Vedolizumab 300 mg, IV infusion, once Q8W that maybe reduced to once Q4W based on the investigator's judgment of participant's clinical status and acknowledged by the medical monitor for up to 6 years.
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 331
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (12.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147
  Male | 184
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 36
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 292
  More than one race | 0
  Unknown or Not Reported | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 13
  Bulgaria | 4
  Czech Republic | 115
  Estonia | 4
  Hungary | 46
  India | 13
  Italy | 5
  Korea, Republic of | 21
  Latvia | 1
  Malaysia | 1
  New Zealand | 6
  Poland | 41
  Romania | 3
  Russian Federation | 35
  Serbia | 1
  Turkey | 5
  Ukraine | 5
  South Africa | 12
Weight [Mean (Standard Deviation); unit: kilograms (kg)] — Population: Number analyzed is the number of participants with data available for weight at Baseline.
  kilograms (kg)
    number analyzed (Participants) | 330
    (all) | 76.91 (16.988)
Height [Mean (Standard Deviation); unit: centimeters (cm)] — Population: Number analyzed is the number of participants with data available for height at Baseline.
  centimeters (cm)
    number analyzed (Participants) | 330
    (all) | 171.4 (11.06)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)] — BMI = weight (kg) / [height (m^2)] Population: Number analyzed is the number of participants with data available for BMI at Baseline.
  kilograms per meter square (kg/m^2)
    number analyzed (Participants) | 330
    (all) | 26.16 (5.667)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the study drug. A SAE is defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires participant hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly/birth defect or is an important medical event. Percentages are rounded off to the nearest decimal point.
Time Frame: From first dose of study drug in this XAP study through 18 weeks after the last dose of study drug (up to 6.3 years)
Population: FAS consisted of all participants enrolled in the XAP study, who received at least 1 dose of study drug (i.e., vedolizumab IV treatment), including the dose given at T0 (last vedolizumab dose in the qualifying study).
Measure: Number; unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 331
percentage of participants
  AEs | 61.9
  SAEs | 15.1

2. Primary Outcome: Percentage of Participants With Adverse Events of Special Interest (AESIs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the study drug. AESIs included serious infections (opportunistic infections, such as progressive multifocal leukoencephalopathy [PML]), malignancies, liver injury, infusion-related hypersensitivity reactions, and injection site reactions. Percentages are rounded off to the nearest decimal point.
Time Frame: From first dose of study drug in this XAP study through 18 weeks after the last dose of study drug (up to 6.3 years)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 331
percentage of participants | 3.9

ADVERSE EVENTS:
Time Frame: From first dose of study drug in this XAP study through 18 weeks after the last dose of study drug (up to 6.3 years)
Description: FAS consisted of all participants enrolled in the XAP study, who received at least 1 dose of study drug (i.e., vedolizumab IV treatment), including the dose given at T0 (last vedolizumab dose in the qualifying study).
Arm/Group | Vedolizumab 300 mg
All-Cause Mortality (participants affected / at risk) | 1/331
Serious Adverse Events (participants affected / at risk) | 50/331
Other Adverse Events (participants affected / at risk) | 100/331
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Vedolizumab 300 mg (N=331)
Abdominal abscess (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amylase increased (Investigations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Anal abscess (Infections and infestations) | 1
Anal fistula (Gastrointestinal disorders) | 1
COVID-19 (Infections and infestations) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Cataract (Eye disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 4/142 — The number affected are the number of participants with preferred disease condition of ulcerative colitis.
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Crohn's disease (Gastrointestinal disorders) | 5/189 — The number affected are the number of participants with preferred disease condition of Crohn's disease.
Device dislocation (Product Issues) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Fracture displacement (Injury, poisoning and procedural complications) | 1
Gastrointestinal viral infection (Infections and infestations) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Goitre (Endocrine disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1
Hypertension (Vascular disorders) | 1
Ileal stenosis (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 2
Large intestinal obstruction (Gastrointestinal disorders) | 1
Large intestinal stenosis (Gastrointestinal disorders) | 1
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myocardial infarction (Cardiac disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Ovarian cyst (Reproductive system and breast disorders) | 1
Peripheral artery dissection (Vascular disorders) | 1
Pneumonia (Infections and infestations) | 1
Pseudopolyposis (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 2
Tibia fracture (Injury, poisoning and procedural complications) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Venous aneurysm (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Vedolizumab 300 mg (N=331)
COVID-19 (Infections and infestations) | 17
Colitis ulcerative (Gastrointestinal disorders) | 20/142 — The number affected are the number of participants with preferred disease condition of ulcerative colitis.
Crohn's disease (Gastrointestinal disorders) | 35/189 — The number affected are the number of participants with preferred disease condition of Crohn's disease.
Hypertension (Vascular disorders) | 21
Nasopharyngitis (Infections and infestations) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT02743806/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT02743806/SAP_001.pdf